CLINICAL TRIAL: NCT07397338
Title: A Phase 1/2 Open-Label, Multicenter Study of RAS(ON) Inhibitors in Combination With Ivonescimab With or Without Other Anti-Cancer Agents in Patients With Solid Tumors
Brief Title: Study of RAS(ON) Inhibitors in Combination With Ivonescimab in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-APEX-103
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors; Non-small Cell Lung Cancer (NSCLC); NSCLC; Colorectal Cancer (CRC); CRC
Keywords: Advanced Solid Tumors; Metastatic Solid Tumors; Non-small Cell Lung Cancer; NSCLC; Colorectal Cancer; CRC; RAS; NRAS; KRAS; HRAS; RAS Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — Carboplatin; Cisplatin; Pemetrexed; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Daraxonrasib + Ivonescimab Combination (Experimental): Dose Exploration and Dose Expansion (+ Carboplatin/Cisplatin + Pemetrexed)
  Interventions: Drug: Daraxonrasib; Drug: Ivonescimab; Drug: Carboplatin/Cisplatin + Pemetrexed (Dose Expansion Only)
- Arm B: Elironrasib + Ivonescimab Combination (Experimental): Dose Exploration and Dose Expansion. Dose Expansion will include two separate cohorts: Cohort B1 (+ daraxonrasib) and Cohort B2 (+ Carboplatin/Cisplatin + Pemetrexed).
  Interventions: Drug: Elironrasib; Drug: Ivonescimab; Drug: Carboplatin/Cisplatin + Pemetrexed (Cohort B2 Only); Drug: Daraxonrasib (Cohort B1 only)
- Arm C: Zoldonrasib + Ivonescimab Combination (Experimental): Dose Exploration and Dose Expansion. Dose Expansion will include two separate cohorts: Cohort C1 and Cohort C2 (+ Cetuximab).
  Interventions: Drug: Zoldonrasib; Drug: Ivonescimab; Drug: cetuximab (Cohort C2 Only)

INTERVENTIONS:
Drug: Daraxonrasib — oral tablets
  Arms: Arm A: Daraxonrasib + Ivonescimab Combination
Drug: Elironrasib — oral tablets
  Arms: Arm B: Elironrasib + Ivonescimab Combination
Drug: Zoldonrasib — oral tablets
  Arms: Arm C: Zoldonrasib + Ivonescimab Combination
Drug: Ivonescimab — IV infusion
Drug: Carboplatin/Cisplatin + Pemetrexed (Dose Expansion Only) — IV infusion
  Arms: Arm A: Daraxonrasib + Ivonescimab Combination
Drug: cetuximab (Cohort C2 Only) — IV infusion
  Arms: Arm C: Zoldonrasib + Ivonescimab Combination
Drug: Carboplatin/Cisplatin + Pemetrexed (Cohort B2 Only) — IV infusion
  Arms: Arm B: Elironrasib + Ivonescimab Combination
Drug: Daraxonrasib (Cohort B1 only) — oral tablets
  Arms: Arm B: Elironrasib + Ivonescimab Combination

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of RAS(ON) inhibitors in combination with ivonescimab in adults with advanced or metastatic solid tumors with a RAS mutation.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/2 study of RAS(ON) inhibitors in combination with ivonescimab with or without other anti-cancer agents in adults with advanced or metastatic solid tumors with a RAS mutation to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary clinical activity. The study consists of three arms: Arm A:daraxonrasib in combination with ivonescimab; Arm B: elironrasib in combination with ivonescimab; and Arm C: zoldonrasib in combination with ivonescimab. All arms consist of two parts: Part 1- dose exploration and Part 2- dose expansion. Part 1 dose exploration will explore the safety and tolerability of individual RAS(ON) inhibitors in combination with ivonescimab. Part 2 dose expansion will explore the safety, tolerability, and antitumor activity of the individual RAS(ON) inhibitors with ivonescimab +/- anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and has provided informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Histologically confirmed, locally advanced or metastatic solid tumor malignancy with documented RAS mutation in KRAS, HRAS, or NRAS.
* Received and progressed or been intolerant to prior standard therapy (Part 1 Dose Exploration).
* Non-squamous NSCLC without a treatable driver mutation in other oncogenes that has not received prior systemic treatment (Arms A & B for Part 2 Dose Expansion).
* Solid tumor or CRC previously treated with no more than 2 prior lines of therapy for advanced disease and progressed or been intolerant to prior standard therapies (Arm C for Part 2 Dose Expansion).
* Measurable disease per RECIST v1.1
* Adequate organ function (bone marrow, liver, kidney, coagulation, endocrine).
* Able to take oral medications.

Exclusion Criteria:

* Head and neck squamous cell carcinoma.
* Any conditions that may affect the ability to take or absorb study drug.
* Major surgery within 4 weeks prior to receiving study drug(s).
* Patient is unable or unwilling to comply with protocol-required study visits or procedures.
* Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) | Up to approximately 4 years
  Number of patients with AEs as assessed by CTCAE v5.
Changes in vital signs | Up to approximately 4 years
  Number of patients with changes in vital signs.
Changes in clinical laboratory test values | Up to approximately 4 years
  Number of patients with changes in clinical laboratory test values.
Dose Limiting Toxicities | 28 days
  Number of patients with dose limiting toxicities

SECONDARY OUTCOMES:
Concentration of RAS(ON) inhibitors and ivonescimab | Up to Cycle 6 Day 1 (each cycle is 21 days)
  Trough and peak blood concentrations of RAS(ON) inhibitors and ivonescimab over time as applicable.
Objective Response Rate (ORR) | Up to approximately 4 years
  ORR per response evaluation criteria in solid tumors (RECIST) v1.1
Duration of Response (DOR) | Up to approximately 4 years
  DOR per RECIST v1.1
Disease Control Rate (DCR) | Up to approximately 4 years
  DCR per RECIST v1.1
Time to response (TTR) | Up to approximately 4 years
  TTR per RECIST v1.1
Progression free survival (PFS) | Up to approximately 4 years
  PFS per RECIST v1.1
Anti-drug Antibody (ADA) of ivonescimab | Up to approximately 4 years
  Number and percentage of patients with anti-ivonescimab antibody

CONTACTS AND LOCATIONS:
Locations (1):
- NEXT Virginia, Fairfax, Virginia, United States